CLINICAL TRIAL: NCT01266317
Title: Open-Label, Feasibility Study of Combined Plasma Exchange (PEX), Rituximab, and Corticosteroids in Patients With Acute Idiopathic Pulmonary Fibrosis Exacerbations
Brief Title: Combined PEX, Rituximab and Steroids in Acute Idiopathic Pulmonary Fibrosis Exacerbations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael Donahoe (Other)
Responsible Party: Sponsor-Investigator, Michael Donahoe, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO10110151
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: IPF
MeSH Terms: interventions — PHEX Phosphate Regulating Neutral Endopeptidase; Rituximab; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined PEX, Rituximab and Steroids (Experimental): Standard Steroid Treatment: One gm of methylprednisolone I.V., on day 0, followed by 40 mg/day I.V. on days 1-4, and days 6-12 (or the P.O. prednisone equivalent). Methylprednisolone 100 mg I.V. will be administered on days 5 and 13. Steroid doses will then be 20 mg methylprednisolone I.V. (or P.O. prednisone equivalent) from days 14-28, and then reduced thereafter at the discretion of the principle investigator.
  Plasma exchange (PEX) will consist of 1.5x estimated plasma volume exchanges for 3 successive days (0, 1,2) and then, after a one day interval to enable equilibration of autoantibodies sequestered in tissues, two more daily treatments on days 4 and 5.
  Rituximab: One gm I.V. will be administered on day 5 (after completion of the last PEX) and day 13.
  Interventions: Drug: Combined Plasma Exchange (PEX), Rituximab, and Corticosteroids

INTERVENTIONS:
Drug: Combined Plasma Exchange (PEX), Rituximab, and Corticosteroids — Standard Steroid Treatment, Plasma exchange will consist of 1.5x estimated plasma volume exchanges, Rituximab

SUMMARY:
This is an open-label Phase I/II trial to assess the feasibility and safety of combined plasma exchange (PEX), rituximab, and conventional corticosteroid administration on the outcome of hospitalized patients with acute IPF exacerbations. The specific aims of this study are:

1. To assess the feasibility and safety of combined PEX, rituximab, and conventional corticosteroid administrations for the treatment of hospitalized patients with acute IPF exacerbations by monitoring indices of respiratory (PaO2) and cardiovascular function during the treatment interval.
2. To assess the efficacy of combined PEX, rituximab, and conventional corticosteroid administrations for the treatment of hospitalized patients with acute IPF exacerbations on patient survival in comparison to historical controls. Patient survival for this investigation will be defined using the composite outcome of 60 day survival and/or survival to lung transplantation.

Subjects between 18 and 80 years of age who have a confirmed diagnosis of IPF, and meet all the study requirements will be enrolled in this study. A total of 10 subjects of both genders and all ethnic backgrounds with acute IPF exacerbations hospitalized at University of Pittsburgh Medical Center will be enrolled in this study.

DETAILED DESCRIPTION:
This is a prospective, open-label Phase II, non-randomized clinical trial to assess the feasibility and safety of combined plasma exchange (PEX), rituximab, and conventional corticosteroid administration in patients with acute IPF exacerbations.

INCLUSION CRITERIA:

1. A diagnosis of idiopathic pulmonary fibrosis that fulfills American Thoracic Society Consensus Criteria.
2. Unexplained worsening or development of dyspnea or hypoxemia within 30 days leading to the current hospitalization.
3. Radiographic imaging showing ground-glass abnormality and/or consolidation superimposed on a background of reticular or honeycomb pattern consistent with UIP.
4. Intent on the part of the treating physician to use high dose steroid therapy as a therapeutic effort to treat a diagnosis of acute IPF exacerbation.

EXCLUSION CRITERIA

1. Diagnosis of documented infection based upon clinical evaluation and microbial testing.
2. Diagnosis of thromboembolic disease by clinical assessment.
3. Diagnosis of an additional etiology for ALI/ARDS based upon clinical assessment to include sepsis, aspiration, trauma, inhalational injury, acute pancreatitis, drug toxicity, blood product transfusion reaction, or stem cell transplantation.
4. Diagnosis of congestive heart failure that accounts for the hypoxemia.
5. Presence of active hepatitis B infection.
6. Coagulopathy defined as an INR > 1.8, PTT > 2 x control, and platelet count < 50K.
7. Hyperosmolar state or diabetic ketoacidosis to suggest uncontrolled diabetes mellitus or uncontrolled hypertension (systolic BP > 160 mm Hg and diastolic BP > 100 mm Hg) which would contraindicated the use of corticosteroids.
8. Hemodynamic instability defined as a vasopressor requirement which would contraindicate the use of plasmapheresis.
9. History of reaction to blood products, murine-derived products, or prior exposures to human-murine chimeric antibodies,
10. History of malignancy.
11. Inability or unwillingness to accept a blood transfusion.
12. Inability or unwillingness to complete post- treatment surveillance for 60 days.
13. Diagnosis of major comorbidities expected to interfere with subjects study participation for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic pulmonary fibrosis that fulfills American Thoracic Society Consensus Criteria.
* Unexplained worsening or development of dyspnea or hypoxemia within 30 days leading to the current hospitalization.
* Radiographic imaging showing ground-glass abnormality and/or consolidation superimposed on a background of reticular or honeycomb pattern consistent with usual interstitial pneumonia.
* Intent on the part of the treating physician to use high dose steroid therapy as a therapeutic effort to treat a diagnosis of acute IPF exacerbation.

Exclusion Criteria:

* Diagnosis of documented infection based upon clinical evaluation and microbial testing.
* Diagnosis of thromboembolic disease by clinical assessment.
* Diagnosis of an additional etiology for Acute Lung Injury/Acute Respiratory Distress Syndrome based upon clinical assessment to include sepsis, aspiration, trauma, inhalational injury, acute pancreatitis, drug toxicity, blood product transfusion reaction, or stem cell transplantation.
* Diagnosis of congestive heart failure that accounts for the hypoxemia.
* Presence of active hepatitis B infection.
* Coagulopathy defined as an International Normalized Ratio > 1.8, Partial Thromboplastin Time > 2 x control, and platelet count < 50,000.
* Hyperosmolar state or diabetic ketoacidosis to suggest uncontrolled diabetes mellitus or uncontrolled hypertension (systolic BP > 160 mm Hg and diastolic BP > 100 mm Hg) which would contraindicated the use of corticosteroids.
* Hemodynamic instability defined as a vasopressor requirement which would contraindicate the use of plasmapheresis.
* History of reaction to blood products, murine-derived products, or prior exposures to human-murine chimeric antibodies,
* History of malignancy.
* Inability or unwillingness to accept a blood transfusion.
* Inability or unwillingness to complete post- treatment surveillance for 60 days.
* Diagnosis of major comorbidities expected to interfere with subjects study participation for 60 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donahoe, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Donahoe M, Valentine VG, Chien N, Gibson KF, Raval JS, Saul M, Xue J, Zhang Y, Duncan SR. Autoantibody-Targeted Treatments for Acute Exacerbations of Idiopathic Pulmonary Fibrosis. PLoS One. 2015 Jun 17;10(6):e0127771. doi: 10.1371/journal.pone.0127771. eCollection 2015. PMID 26083430

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined PEX, Rituximab and Steroids: Standard Steroid Treatment: One gm of methylprednisolone I.V., on day 0, followed by 40 mg/day I.V. on days 1-4, and days 6-12 (or the P.O. prednisone equivalent). Methylprednisolone 100 mg I.V. will be administered on days 5 and 13. Steroid doses will then be 20 mg methylprednisolone I.V. (or P.O. prednisone equivalent) from days 14-28, and then reduced thereafter at the discretion of the principle investigator.
  Plasma exchange (PEX) will consist of 1.5x estimated plasma volume exchanges for 3 successive days (0, 1,2) and then, after a one day interval to enable equilibration of autoantibodies sequestered in tissues, two more daily treatments on days 4 and 5.
  Rituximab: One gm I.V. will be administered on day 5 (after completion of the last PEX) and day 13.
  Combined Plasma Exchange (PEX), Rituximab, and Corticosteroids: Standard Steroid Treatment, Plasma exchange will consist of 1.5x estimated plasma volume exchanges, Rituximab
Period: Overall Study
Arm/Group | Combined PEX, Rituximab and Steroids
Started | 9 (One additional patient was a protocol violation post consent when autoantibodies returned positive)
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Combined PEX, Rituximab and Steroids
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory and/or Hemodynamic Deteriorations
Description: To assess the feasibility and safety of combined PEX, rituximab, and conventional corticosteroid administrations for the treatment of hospitalized patients with acute IPF exacerbations by monitoring indices of respiratory (PaO2) and cardiovascular function during the treatment interval. Respiratory deterioration was defined by a compilations of respiratory deteriorations (deteriorating gas exchange) and hemodynamic deteriorations (defined as a need for medical intervention).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PEX, Rituximab and Steroids
Number analyzed (Participants) | 7
Participants
  Respiratory Deterioration | 1
  Hemodynamic Deterioration | 3

2. Secondary Outcome: Number of Participants Survived to 60 Days or to Transplantation
Description: The secondary outcome measures a composite outcome defined as survival to 60 days or survival to transplantation at any time post therapy.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PEX, Rituximab and Steroids
Number analyzed (Participants) | 7
Participants | 3

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Combined PEX, Rituximab and Steroids
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined PEX, Rituximab and Steroids (N=10)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject underwent dialysis catheter placement for plasmapheresis and had a marked desaturation at the conclusion of the procedure. Subject was intubated due to hypoxemia. The study treatment was withheld until the subject has been stabilized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined PEX, Rituximab and Steroids (N=10)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Infection (Skin and subcutaneous tissue disorders) | 1 (1) — Catheter infection

LIMITATIONS AND CAVEATS:
This was a pilot, open-label trial of an unprecedented regimen for a highly lethal disease and, as such, included only small numbers of subjects and historical controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes